CLINICAL TRIAL: NCT05829759
Title: Brothers Building Brothers by Breaking Barriers for Telehealth Delivery (Tele-B6)
Brief Title: Telehealth Delivery (Tele-B6)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sophia Hussen, Associate Professor of Public Health and Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003404; R34MH129187-01 (NIH); 2025P013132 (Other: Emory IRB)
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: HIV Seropositivity; Bisexuality
Keywords: black; Multiracial identity
MeSH Terms: conditions — HIV Seropositivity; Bisexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-B6 (Experimental): The tele-B6 intervention includes six group sessions delivered over the course of six weeks. Survey assessments for the intervention group will be conducted at enrollment (baseline), 2 months (immediate post-intervention survey), 4 months (interim-survey, post-intervention), and 6 months (endline).
  Interventions: Behavioral: Tele-B6
- Wait-list control -delayed intervention (Other): Await-list control design to safeguard ethical treatment of participants by ensuring that a potentially impactful intervention will be available to all after a brief waiting period.
  Interventions: Behavioral: Delayed intervention (waitlist control)

INTERVENTIONS:
Behavioral: Tele-B6 — Participants will be part of the Tele-B6 intervention that includes six group sessions delivered over the course of six weeks. Survey assessments for the intervention group (first phase) will be conducted at enrollment (baseline), 2 months (immediate post-intervention survey), 4 months (interim-survey, post-intervention), and 6 months (endline).
  Arms: Tele-B6
Behavioral: Delayed intervention (waitlist control) — Wait-list control participants will be assigned to a group for initiation of the full intervention beginning at month 4 after their enrollment (i.e., beginning after they, and their corresponding intervention group, have completed their intervention and two follow-up surveys). Wait-list control participants will complete surveys at enrollment (baseline), 2 months (pre-intervention), 4 months (preintervention), 6 months (immediate post-intervention), and 8 months (post-intervention).
  Arms: Wait-list control -delayed intervention

SUMMARY:
The research team has developed an interventional group program for young men living with HIV and will be adapting it for telehealth delivery. The purpose of the study is to determine whether or not this program can help improve social connections and the health of young men in online delivery and evaluate its potential for implementation in a community setting. The study has three phases: (1) engaging a community advisory board to create and adapt the intervention for online delivery, (2) a randomized clinical trial of the online intervention, and (3) evaluation of the program for community implementation with our partner organization. Participants in the second phase of the study will meet with a study team member to discuss the research process and provide informed consent. The community organization employees will provide consent online prior to completion of a survey and indicate whether they consent to be contacted further for in-depth interviews.

DETAILED DESCRIPTION:
Subjects will participate in synchronous, online discussion sessions via videoconference for two hours per week over a six-week period. Sessions will include engaging educational components and interactive activities including discussions of case scenarios and sharing of personal experiences where desired. At the end of each videoconference session, participants will be asked to complete a brief session evaluation form in which they will rate the content, facilitation, and overall experience for the week. The long-term goal is to improve engagement across the HIV continuum of care (HIV-CoC) by enhancing individual- and community-level resilience processes among young Black gay, bisexual and other men who have sex with men (YB-GBMSM) living with HIV. To this end, the research team has used community-based participatory research methods to develop Brothers Building Brothers by Breaking Barriers (B6), a novel group-level intervention designed to affirm intersectional identities and augment social capital among YB-GBMSM. The goal of this current study is to adapt and pilot B6 for telehealth delivery (creating tele-B6) within the context of an established community-based organization (CBO), as a strategy for enhancing feasibility and scalability prior to a larger efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Black race, inclusive of multiracial identities; male gender, inclusive of transgender men;
* self-identification as gay, bisexual, or another non-heterosexual orientation, and/or any history of consensual anal or oral sex with men;
* HIV-positive serostatus;
* age 18-29 years inclusive;
* residence in the Atlanta Metropolitan Statistical Area;
* available and interested to meet for two hours weekly over a six-week period.

Exclusion Criteria:

* Age < 18 years or > 30 years
* Unwilling or unable to provide written informed consent
* Enrollment in one phase of the study is an exclusion criterion for enrollment in other phases

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — male gender, inclusive of transgender men
Enrollment: 60 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Acceptability | Study Exit (up to 8* months)
  Qualitative interviews: Open-ended questions adapted from the original B6 exit interview guide.
  *8-month timepoint only applies to waitlist control participants
Change in the Acceptability Surveys | 2, 4, 6, up to 8* months
  Post-session evaluation forms (adapted from original B6) after each group session.
  *8-month timepoint only applies to waitlist control participants
Change in Recruitment Rates | 2, 4, 6, up to 8* months
  Rates of participation from screened and eligible participants.
  *8-month timepoint only applies to waitlist control participants
Change in retention | 2, 4, 6, up to 8* months
  Attendance logs during each visit.
  *8-month timepoint only applies to waitlist control participants
Change in the intervention fidelity | 2, 4, 6, up to 8* months
  Review of the Structured intervention logs (adapted from original B6)
  *8-month timepoint only applies to waitlist control participants
Safety (adverse events) | During study participation up to 8* months
  Review of Adverse event tracking forms
  *8-month timepoint only applies to waitlist control participants

SECONDARY OUTCOMES:
Change in Perception of Structural Racism and Discrimination. | 0, 2, 4, 6, 8* months
  Participants will complete surveys measuring socioeconomic status, material resources scale. The material resources survey has 18 questions asking how often the participants' family needs are adequately met. There are six options (never=0; rarely=1; less than half of the time=w, about half of the time=3; more than half of the time=4; and always=5). The highest score means that needs are adequately met.
  *8-month timepoint only applies to waitlist control participants
Change in Perception of discrimination | 0, 2, 4, 6, up to 8* months
  Participants will complete the Everyday Discrimination Scale at baseline and after each session. Each response is given a value according to the Likert scale ('never'=1 to 'almost everyday'=6). Responses are summed across items to produce a score ranging from 10 to 60. A higher score may indicate higher perception of discrimination.
  *8-month timepoint only applies to waitlist control participants
Change in Perception of HIV stigma | 0, 2, 4, 6, up to 8* months
  Participants will complete the HIV stigma scale at baseline and after each session. This scale includes which includes 10 item stigma rated on a 5-point scale from "Strongly Disagree" to "Strongly Agree".
  *8-month timepoint only applies to waitlist control participants
Change in Perception of internalized homonegativity inventory | 0, 2, 4, 6, up to 8* months
  Participants will complete the internalized homonegativity inventory at baseline and after each session.
  This 26-item scale has four subscales: (a) Public Identification as Gay, (b) Perception of Stigma Associated with Being Gay, (c) Social Comfort with Gay Men, (d) Moral and Religious Acceptability of Being Gay.
  *8-month timepoint only applies to waitlist control participants
Qualitative description of intersectional stigma | Exit of study (up to 8 months)
  Participants will be asked to complete surveys with open-ended questions adapted from the original B6 exit interview guide. There is no summary score of the open-ended questions asked during the interview.
  *8-month timepoint only applies to waitlist control participants
Change in intersectional stigma | Exit of study (up to 8 months)
  Participants will be asked to complete surveys with open-ended questions adapted from the original B6 exit interview guide. There is no summary score of the open-ended questions asked during the interview.
  *8-month timepoint only applies to waitlist control participants
Change in logistical barriers | 0, 2, 4, 6, up to 8* months
  Participants will be asked to complete surveys and matched to Zipcode to derive neighborhood measures.
  *8-month timepoint only applies to waitlist control participants
Qualitative description of logistical barriers | Exit of study (up to 8 months)
  Participants will be asked to complete open-ended questions adapted from the original B6 exit interview guide. There is no summary score of the open-ended questions asked during the interview.
  *8-month timepoint only applies to waitlist control participants
Changes in perception of individual resilience process: Identity Affirmation | 0, 2, 4, 6, up to 8* months
  Participants will complete the multidimensional model of black identity lesbian, gay, and bisexual identity scale,
  *8-month timepoint only applies to waitlist control participants
Qualitative description individual resilience process: Identity Affirmation | Exit of study (up to 8 months)
  Participants will be asked to complete open-ended questions adapted from the original B6 exit interview guide. There is no summary score of the open-ended questions asked during the interview.
  *8-month timepoint only applies to waitlist control participants
Changes in the community resilience process: social capital | 0, 2, 4, 6, up to 8* months
  Participants will complete the personal social capital scale. A five-point Likert scale is used to assess these questions with 1 = none and 5 = all. A composite score will be derived by summarizing the item scores such that a higher score indicates a greater perceived collective efficacy.
  *8-month timepoint only applies to waitlist control participants
Qualitative description of the community resilience process: social capital | Exit of study (up to 8 months)
  Participants will be asked to complete open-ended questions adapted from the original B6 exit interview guide. There is no summary score of the open-ended questions asked during the interview.
  *8-month timepoint only applies to waitlist control participants
Changes in the perception of minority stress: depression | 0, 2, 4, 6, up to 8* months
  Participants will complete the Studies Depression Scale (CES-D) survey. In scoring the CES-D, a value of 0, 1, 2, or 3 is assigned to a response depending upon whether the item is worded positively or negatively. The possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology.
  *8-month timepoint only applies to waitlist control participants
Changes in the perception of minority stress: general well-being | 0, 2, 4, 6, up to 8* months
  Participants will complete the general well-being (GWB) survey. The General Well-Being Schedule (GWB) is designed to assess an individual's mental health or quality of life. The GWB consists of 18 items indicating subjective feelings of psychological well-being and distress. All of the items utilize the past month as the time frame of interest. The first 14 questions use a six-point rating scale that represents either intensity or frequency. The remaining items use a 0-10 rating scale that is anchored by adjectives. Because some items are reverse scored (items 1, 3, 6, 7, 9, 11, 15, and 16), 14 is subtracted from the total score, yielding a total possible range of scores from 0 to 110. Low scores represent greater distress. Proposed cutoffs representing three levels of distress are 0-60 (severe distress), 61-72 (moderate distress), and 73-110 (positive well-being).
  *8-month timepoint only applies to waitlist control participants
Qualitative description of the minority stress | Exit of study (up to 8 months)
  Participants will be asked to complete open-ended questions adapted from the original B6 exit interview guide. There is no summary score of the open-ended questions asked during the interview.
  *8-month timepoint only applies to waitlist control participants

OTHER OUTCOMES:
Changes in HIV viral load | 0 and 6 months
  The research team will review the electronic medical record (EMR) to abstract HIV viral load information
Rate of retention care | 0 and 6 months
  The research team will review the electronic medical record (EMR) to abstract data on missed appointments

CONTACTS AND LOCATIONS:
Overall Officials: Sophia A. Hussen, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Grady Infectious Diseases Program Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share the results of surveys and clinical abstracted data in a de-identified dataset.
Time Frame: The de-identified dataset will be available after the study and data analysis are complete.
Access Criteria: All requests should be sent by email to the principal investigator.

REFERENCES:
- [Derived] Reed MO, Bullock M, Newman A Jr, Dutta S, Opara SCO, Tewodros T, Doraivelu K, Camacho-Gonzalez A, Murden R, Gamarel K, Harper GW, Hussen SA. Brothers Building Brothers by Breaking Barriers: Protocol for a Pilot Trial of a Telehealth Social Capital Intervention for Young Black Sexual Minority Men Living With HIV. JMIR Res Protoc. 2025 Dec 1;14:e69961. doi: 10.2196/69961. PMID 41325601

DOCUMENTS (1):
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT05829759/ICF_000.pdf